CLINICAL TRIAL: NCT03319576
Title: Early Feeding Following Percutaneous Gastrostomy Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1074
Record Dates: First submitted 2017-09-25; First posted 2017-10-24 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Gastrostomy
Keywords: Gastrostomy; Feeding; G-tube

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early feeding (Experimental): Patients randomized to early feeding will be fed 4 hours following gastrostomy tube placement
  Interventions: Other: Feeding at 4 hours
- Standard feeding (No Intervention): Patients randomized to standard feeding will be fed 24 hours following gastrostomy tube placement

INTERVENTIONS:
Other: Feeding at 4 hours — Patients will be fed 4 hours after their gastrostomy tube placement procedure.
  Arms: Early feeding

SUMMARY:
This study plans to learn more about the safety of early feeding following placement of a feeding tube. Doctors in other specialties feed patients 4 hours after patients receive a feeding tube. However, Interventional Radiologists typically wait to feed patients for 24 hours following feeding tube placement. The investigator would like to demonstrate that feeding after 4 hours does not increase complications and can actually reduce the burden to patients who receive a feeding tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-80 years
* Outpatients receiving a gastrostomy tube at University of Colorado that do not require post-pyloric feeding
* Patients that have no contraindication for intragastric feeding immediately following tube placement
* INR (international normalized ratio) <1.5
* Platelet count > 50,000/µL
* WBC (white blood cell count) 4.0-11.1 x 109/L

Exclusion Criteria:

* Patients < 18 years or > 80 years of age
* Patients admitted to the hospital at the time of screening (i.e., inpatients)
* Women who are pregnant (confirmed by urine pregnancy screen)
* Patients requiring post-pyloric feeding
* Patients receiving venting gastrostomy tubes
* Patients receiving primary Gastro-Jejunal (GJ) Tube tube placement
* Patients with an interposed bowel on CT after stomach insufflation
* INR > 1.5
* Platelet count < 50,000/µL
* WBC > 11.1 x 109/L
* Known active infection
* Need for post-gastric feeding
* History of gastric bypass surgery or Roux-En-Y
* Mechanical obstruction of the GI tract
* Active peritonitis
* Known hemodynamic instability as demonstrated by tachycardia, hypotension, labile blood pressure or altered mental status.
* Bowel ischemia
* Ascites
* Recent Gastro-Intestinal (GI) bleeding (within 2 weeks)
* Respiratory compromise as demonstrated by hypercarbia (CO2>45mmHg) or hypoxia (O2<90%)
* Unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Inability to feed | 4 hours after gastrostomy tube placement
  Inability to feed due to high pre-feeding gastric residual volume
Changes in any major or minor complications | 24 hours after gastrostomy tube placement
  Any change(s) noted in any major and/or minor complications arising post gastrostomy tube placement will be evaluated.

SECONDARY OUTCOMES:
Positive predictive value of computed tomography (CT) prior to gastrostomy tube placement will be measured at the end of the study. | At Study Completion, approximately 2 years
  Positive predictive value of CT prior to gastrostomy tube placement
Procedural experience from the patients' perspective | 2 weeks after gastrostomy tube placement
  Patients will be asked to complete a survey related to tube usage and difficulties with feeding and immediate post-procedural complications

CONTACTS AND LOCATIONS:
Overall Officials: Premal Trivedi, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data outside of the study team.